CLINICAL TRIAL: NCT05793619
Title: Evaluation of the Tolerance and Performance (Mode of Administration) of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots
Brief Title: Tolerance and Performance (Mode of Administration) of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry); CEISO (Industry); LTD HEALTH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_8
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-06

CONDITIONS: Lentigo Solar; Senile Lentigo
Keywords: cryotherapy; hyperpigmentation; Skin Diseases
MeSH Terms: conditions — Hyperpigmentation; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1 : prototypes (816-v1 301) to (816-v1 355) every week (Experimental): Application on the brown spots of the face for the prototypes (816-v1 301) to (816-v1 355) at D0, D7, D14, D21, D28 and D35
  Interventions: Device: Prototypes (816-v1 301) to (816-v1 355) every week
- Condition 2 : prototypes (816-v1 301) to (816-v1 355) every two weeks (Experimental): Application on the brown spots of the face for the prototypes (816-v1 301) to (816-v1 355) at D0, D14, D28, D42, D56 and D70
  Interventions: Device: Prototypes (816-v1 301) to (816-v1 355) every two weeks

INTERVENTIONS:
Device: Prototypes (816-v1 301) to (816-v1 355) every week — Application on brown spots located on the face (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face. Subjects will be lying down, and the prototypes will be administered upside down. During applications, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 1 : prototypes (816-v1 301) to (816-v1 355) every week
Device: Prototypes (816-v1 301) to (816-v1 355) every two weeks — Application on brown spots located on the face (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face. Subjects will be lying down, and the prototypes will be administered upside down. During applications, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 2 : prototypes (816-v1 301) to (816-v1 355) every two weeks

SUMMARY:
CS5_8 study aim to evaluate the tolerance and to adjust the mode of administration of 2 different conditions of cryotherapy treatments applied on the brown spots of the face with 1 prototype (816-v1). Each treatment corresponds to a specific frequency of cryogenic spray application.

The study will evaluate the following prototype :

• Prototypes from (816-v1 301) to (816-v1 355)

DETAILED DESCRIPTION:
Rational :

Solar/senile lentigo is a harmless patch of darkened skin. It results from exposure to ultraviolet (UV) radiation, which causes local proliferation of melanocytes and accumulation of melanin within the skin cells (keratinocytes). Solar/senile lentigos or lentigines are very common, especially in people over the age of 40 years.

Solar/senile lentigines are found as groups of similar lesions on sun-exposed sites, particularly the face or the back of hands.

Cryotherapy is more and more used to improve skin appearance and currently used to treat lentigo spot. However, the cryogenic gas (conventional cryotherapy - liquid nitrogen) creates a dermabrasion of the skin surface and person receiving this kind of treatment presents an impaired skin during a few days following the treatment as temporary damage of stratum corneum, erythema, scars, burns.

Following the side effects occurring after conventional cryotherapy application, the Sponsor has developed some devices using difluoroethane, manufactured by CRYONOVE PHARMA, already available on the local and international markets, e.g. CRYOBEAUTY MAINS and CRYOBEAUTY CORPS.

To continue it research and development activities, the sponsor selected other sequences of a cryogenic spray (1 prototype of devices for face used according to different frequencies of application, i.e. 2 conditions evaluated) which could be used for lentigo treatment with a same benefit for the consumers without any safety outcomes.

Design:

The study performed is a proof of performance designed to be exploratory, interventional study, monocentric, randomized and double blinded.

Intervention :

1 prototype of devices are evaluated in 2 different conditions. Each treatment corresponds to a specific frequency of cryogenic spray application. A total of 42 brown spots are needed (at least 1 brown spot on the face).The 42 brown spots will be randomized between the 2 conditions and will be attributed to subjects according to the number of spots identified by Investigator.

Prototypes (816-v1 301) to (816-v1 355) will be applied on brown pots located on the face. Each spot will be treated six times by a defined prototype (always the same device on the same spot all along the study) according to specific frequencies (every week or every two weeks).

Prior to any study device application, the dermatologist will assess the adverse events and will decide if the period between two consecutive applications should be extended or not.The dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.

As the study will use prototypes, before each treatment, the prototype will be administered to any surface (in order to purge eventually the presence of air). An operator previously trained by the dermatologist will apply the study device to the patient's face.

Subjects will be lying down, and the device will be administered upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.

The patient follow-up visits are from Day 0 to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* Ages 30 to 75.
* Phototypes I to IV (according with Fitzpatrick scale)
* Featuring brown spots (solar lentigos, senile lentigo) on the face ≥ 3 and ≤ 6 mm in diameter (at least 1 spots per subject)
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for their participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, facials, UV ...) in the month before the start of the study, at the level of the face.
* Having applied a depraving product in the month prior to the start of the study, at the level of the face.
* Having performed cosmetic treatments in a dermatologist (laser, Intense Pulse Light, peeling, creams, cryotherapy ...), at the level of the face in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write Georgian language.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman who does not have a contraceptive method.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 6 points (0 to 5) will be used :
  0=Clear of hyperpigmentation;
  1. Almost clear of hyperpigmentation;
  2. mild, but noticeable hyperpigmentation;
  3. moderate hyperpigmentation (medium brown in quality);
  4. severe hyperpigmentation (dark brown in quality);
  5. very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 5 points will be used (0 to 4):
  0=no hypopigmented lesion;
  1. very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin;
  2. slight area of hypopigmentation of small size and slightly fairer than the surrounding skin;
  3. moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin;
  4. severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and surrounded spotless skin area around the spot skin to assess erythema, oedema blister, bubble, scars, micro-bruise, hematoma, dryness,desquamation, fissures/cracks, roughness,crust, pink spots and papules.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Change from baseline skin sensation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and around the spot skin to assess tightness, stinging, itching, warm and burning sensation.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Self-assesment of pain by VAS | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The pain of the treatment will be assessed by the Visual Analogue Scale (VAS) at time T0 on the treated area.
  The pain assessed is that felt during the application of the devices. It will be collected from the patient within 5 minutes of application.
  The VAS is made up of a 10-centimeter line anchored by two ends of the pain. 10 is the first end being the "maximum pain imaginable" and 0 is the other end being "no pain".
Change from baseline spots visibility | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE) which allows realizing high resolution skin pictures. The capture will be taken on the previously selected lentigo and a spotless area.
Change from baseline spots color | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  L'OREAL Color-Chart is a visual mode of evaluation chart which includes 4 items :
  * Color of lentigo spot
  * Lightness of lentigo spot
  * Color of spotless area
  * Lightness of spotless area
  The items color of lentigo spot and color of spotless area are using a scale redder to yellower in 7 points (G to M).
  The items lightness of lentigo spot and lightness of spotless are using a scale lighter to darker in 15 points (5 to 19)
Change from baseline lentigines global improvement scale (LGIS) score | Day 49 and Day 84
  Lentigines Global Improvement Scale (LGIS) score will be used to assess the spots visibility
  This is a 7-point scale :
  * Completely clear - 0 - : No evidence of hyperpigmentation 100% improvement
  * Almost clear - 1 - : Very significant clearance (about 90%); only minor evidence of hyperpigmentation remains
  * Marked improvement - 2 - : Significant improvement (about 75%); score evidence of hyperpigmentation remains
  * Moderate improvement - 3 - : intermediate between marked and slight improvement; about 50% improvement in the appearance of hyperpigmentation
  * Slight improvement - 4 - : some improvement (about 25%); however significant evidence of hyperpigmentation remains
  * No change - 5 - : Hyperpigmentation has not changed since baseline
  * Worse - 6 - : Worse (hyperpigmentation is worse that at baseline)

SECONDARY OUTCOMES:
Self assessment of skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The skin appearance will be assessed by subjects through a 3 items questionnaire.
  It allows obtaining the subjective appraisal of subject on the treatments using the following 5-point scale:
  * agree,
  * quite agree
  * neither agree, nor disagree
  * quite disagree
  * disagree.
  The items are the following:
  * The spot seems clearer.
  * The size of the spot seems reduced.
  * The spot seems less visible.

CONTACTS AND LOCATIONS:
Overall Officials: Lela BERIDZE, Principal Investigator — LTD HEALTH
Locations (1):
- Ltd "Health", Batumi, Georgia

IPD SHARING:
Plan to Share IPD: No